CLINICAL TRIAL: NCT00007800
Title: Obesity Treatment and NIDDM in Black and White Women
Brief Title: NEW DAY: Nutrition, Exercise, Weight Loss, Diabetes And You
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: Smith-West (completed); R01DK054041 (NIH); NCT00331266 (obsolete NCT alias)
Record Dates: First submitted 2001-01-05; First posted 2001-01-05 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: obesity treatment; non insulin dependent diabetes; type 2 diabetes; behavioral weight control; motivational interviewing; motivational enhancement
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Motivational Interviewing

INTERVENTIONS:
Behavioral: Behavioral Group Weight Loss Intervention
Behavioral: Motivational Interviewing

SUMMARY:
This clinical trial examines whether the addition of individual sessions of a motivational intervention to a state-of-the art behavioral group weight loss intervention for overweight women with Type 2 diabetes improves the weight losses and glycemic control outcomes.

DETAILED DESCRIPTION:
The multi-disciplinary behavioral, group-based intervention focuses on dietary and exercise changes, with group meetings over an 18-month period. Participants are assessed at 6-month intervals (for a total of 18 months) to examine the impact of the interventions on body weight and blood sugar control (primary outcomes), as well as on blood pressure, cholesterol, quality of life and attitudes (secondary outcomes). All enrolled participants receive group-based weight loss intervention. Half the women enrolled also receive several individual sessions of motivational interviewing and the other half of enrolled women receive the same number of individual sessions of health education, which focus on issues relevant to women (e.g., mammography, sleep hygiene, menopause, etc).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 27 - 50
* Type 2 diabetes currently treated with oral medications
* Ability to walk for exercise

Exclusion Criteria:

* Use of insulin
* Current pregnancy
* Presence of debilitating disease, psychotic condition or any other condition that might interfere with participation
* Failure to complete self monitoring diary for 1 week
* Plans to move out of the area in the upcoming 18 months

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218
Dates: Start 2000-05; Study Completion 2002-05

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States